CLINICAL TRIAL: NCT00209911
Title: Atrial and Ventricular Volume and Function In Atrial Fibrillation - A Magnetic Resonance Imaging Study
Brief Title: Study of the Effect of Cardioversion on Cardiac Volume in Patients With Persistent Atrial Fibrillation
Status: Terminated | Type: Observational
Sponsor: Hvidovre University Hospital (Other)
Collaborators: The Foundation of 17.12.1981 (Other); AP Moeller Foundation (Other); Danish Hospital Foundation for Medical Research, Region of Copenhagen (Unknown); Danish Heart Foundation (Other); Copenhagen Hospital Corporation (Other)
Other Study IDs: susette_phd
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2005-09-21 (Estimated); Status verified 2001-01

CONDITIONS: Atrial Fibrillation
Keywords: atrial volume; ventricular volume; atrial function; ventricular function; magnetic resonance imaging; cardioversion; natriuretic peptides
MeSH Terms: conditions — Atrial Fibrillation | interventions — Electric Countershock

STUDY DESIGN:
Observational Model: Natural History | Time Perspective: Prospective

INTERVENTIONS:
Procedure: cardioversion

SUMMARY:
The main objectives in this study were to examine the cardiac structural and functional changes in patients with persistent and permanent AF, with the aim of improving our understanding of the underlying pathophysiological mechanisms. In addition we aimed to identify variables predictive of recurrent AF.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* severe pulmonary or renal disease
* contraindications to magnetic resonance imaging
* valvular disease
* previous cardiac surgery

Min Age: 0 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60
Dates: Start 2001-01; Study Completion 2003-01

CONTACTS AND LOCATIONS:
Overall Officials: Susette Krohn Therkelsen, MD, phd, Principal Investigator
Locations (1):
- Dept. of Cardiology, Copenhagen University Hospital Hvidovre, Hvidovre, Denmark

REFERENCES:
- [Background] Therkelsen SK, Groenning BA, Svendsen JH, Jensen GB. Atrial and ventricular volume and function in persistent and permanent atrial fibrillation, a magnetic resonance imaging study. J Cardiovasc Magn Reson. 2005;7(2):465-73. doi: 10.1081/jcmr-200053618. PMID 15881530